CLINICAL TRIAL: NCT03808012
Title: Predictability of the Ability to Perform an Emergency Stop After Surgery for Inguinal Hernia
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Unsuccessful recruitment
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 001/2019BO2
Record Dates: First submitted 2019-01-14; First posted 2019-01-17 (Actual); Last update posted 2020-12-29 (Actual); Status verified 2019-01

CONDITIONS: Inguinal Hernia
MeSH Terms: conditions — Hernia, Inguinal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Braking after inguinal hernia surgery (Experimental): Cohort testing of driving performance in a brake simulator in patients before and after scheduled inguinal hernia surgery
  Interventions: Other: Braking performance in a brake simulator

INTERVENTIONS:
Other: Braking performance in a brake simulator — Braking performance is tested in a real middle size car cabin to simulate ergonomic conditions of driving a car. This testing cabin has been equipped with customised equipment to allow measurement of reaction time, foot transfer time, brake response time and brake force.

SUMMARY:
Several studies exist on patient performance in drive simulators especially around and after surgery. Recommendations concerning the ability to drive after inguinal hernia are scarce and so far do not offer conclusive results. Aim of the study is to analyse reaction time and foot transfer time (together brake response time) and brake force in a brake simulator before and after scheduled inguinal hernia surgery (Liechtenstein procedure).

ELIGIBILITY:
Inclusion Criteria:

* scheduled surgery for inguinal hernia of the right groin with Lichtenstein procedure
* valid driving license
* male and female

Exclusion Criteria:

* lacking driving license
* pregnancy
* neuromuscular disorder (e.g. myopathy, muscular dystrophy)
* central neurological disorders/diseases (e.g. apoplexia, psychiatric diseases)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-04-10 (Actual); Primary Completion 2020-04-09 (Estimated); Study Completion 2020-07-30 (Estimated)

PRIMARY OUTCOMES:
Braking performance 1 | measurements will be: preoperatively, 2 days postoperatively
  Improvement of Braking performance from preoperatively to 2 days postoperatively in the brake simulator with the focus on brake response time (ms)
Braking performance 2 | measurements will be: preoperatively, 8 days postoperatively
  Improvement of Braking performance from preoperatively to 8 days postoperatively in the brake simulator with the focus on brake response time (ms)

CONTACTS AND LOCATIONS:
Overall Officials: Ulf K Hofmann, MD, Principal Investigator — University Hospital Tuebingen
Locations (1):
- University Hospital Tuebingen, Department of Orthopaedics, Tübingen, Germany

IPD SHARING:
Plan to Share IPD: Undecided